CLINICAL TRIAL: NCT07093762
Title: Efficacy and Safety Analysis of First-Line ABCP Four-Drug Combination Therapy in Advanced SMARCA4-Mutated Non-Small Cell Lung Cancer: A Multicenter, Single-Arm, Prespecified Subgroup Clinical Trial
Brief Title: Efficacy and Safety Analysis of First-Line ABCP Therapy in Advanced SMARCA4-Mutated NSCLC
Status: Not yet recruiting | Type: Observational
Sponsor: Fuzhou General Hospital (Other)
Collaborators: 900 Hospital of Joint Logistics Support Force of PLA (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-059
Record Dates: First submitted 2025-06-29; First posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Non Small Cell Lung Cancer
Keywords: SMARCA4; NSCLC; treatment efficacy; biomarker
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Treatment-naive patients with advanced SMARCA4-mutated NSCLC: 1. Patients pathologically confirmed as having NSCLC, with histologically or cytologically confirmed unresectable locally advanced (Stage IIIB/IIIC) that is not amenable to curative-intent concurrent chemoradiotherapy, metastatic, or recurrent (Stage IV) non-squamous NSCLC, staged according to the IASLC 9th Edition Lung Cancer TNM Staging System by the International Association for the Study of Lung Cancer and the Union for International Cancer Control;
  2. Confirmed SMARCA4 mutation (by NGS testing);
  3. ECOG PS 0-1, with no prior systemic therapy;
  4. Absence of driver gene mutations such as EGFR, ALK, or ROS1;
  5. Patients who can provide sufficient blood samples (see sample requirements for details) and complete basic clinical data, including age, gender, smoking history, family history, lesion location(s), lesion size(s), number of lesions, tumor markers, pathological indicators, treatment information, and re-examination/follow-up information;
  6. Voluntary participation wi
  Interventions: Drug: Atezolizumab+Bevacizumab+Carboplatin+Paclitaxel

INTERVENTIONS:
Drug: Atezolizumab+Bevacizumab+Carboplatin+Paclitaxel — Atezolizumab: 1200 mg IV every 3 weeks; Bevacizumab: 15 mg/kg IV every 3 weeks; Carboplatin: AUC 5 IV every 3 weeks; Paclitaxel: 175 mg/m² IV every 3 weeks. Treatment cycles: After 4-6 cycles, continue Atezolizumab + Bevacizumab as maintenance therapy until disease progression or unacceptable toxicity.

SUMMARY:
SMARCA4 mutation is clinically known to be an independent poor prognostic factor. Both TCGA and the investigators institution's preliminary research indicate that the median overall survival (OS) of mutated patients is significantly shorter than that of wild-type patients (32 months vs. 157.7 months, respectively, P=0.001); it is associated with chemotherapy/immunotherapy resistance, rapid progression, and poor prognosis (OS<12 months). Current standard first-line treatments (such as platinum-based chemotherapy ± immunotherapy) have limited efficacy in SMARCA4-mutated patients (ORR<30%, PFS<4 months). Additionally, NapsinA-positive expression can improve the survival of mutated patients (median OS: 32 months vs. 15 months, P=0.033), but this effect exists only in the SMARCA4-mutated group.

The ABCP regimen has a synergistic mechanism: Atezolizumab (anti-PD-L1): reverses the immunosuppressive microenvironment; Bevacizumab (anti-VEGF): inhibits angiogenesis and enhances T-cell infiltration; Platinum + Paclitaxel: directly kill tumor cells and release neoantigens. Therefore, the investigators preset that SMARCA4 mutation may affect chemotherapy/immunotherapy response through epigenetic regulation, and its value as a predictive biomarker needs to be validated. Hence, the purpose of this study is to observe and explore the efficacy and safety of first-line ABCP four-drug combination therapy in patients with advanced SMARCA4-mutated non-small cell lung cancer.

DETAILED DESCRIPTION:
SMARCA4 is the core catalytic subunit of the SWI/SNF chromatin remodeling complex, and its loss-of-function mutations are closely associated with the development of lung cancer and poor prognosis. Studies show that SMARCA4 mutations account for approximately 5-10% of advanced NSCLC, are more common in males and smokers, and have a significantly higher incidence in large cell carcinoma (LCC) than in other histological subtypes (51.4% in LCC). Data from Asian cohorts show that SMARCA4 mutations are mutually exclusive with driver gene mutations such as EGFR and ALK, and are often accompanied by high tumor mutational burden (TMB) and low PD-L1 expression.

SMARCA4 mutation is clinically known to be an independent poor prognostic factor. Both TCGA and the investigators institution's preliminary research indicate that the median overall survival (OS) of mutated patients is significantly shorter than that of wild-type patients (32 months vs. 157.7 months, respectively, P=0.001); it is associated with chemotherapy/immunotherapy resistance, rapid progression, and poor prognosis (OS<12 months). Current standard first-line treatments (such as platinum-based chemotherapy ± immunotherapy) have limited efficacy in SMARCA4-mutated patients (ORR<30%, PFS<4 months). Additionally, NapsinA-positive expression can improve the survival of mutated patients (median OS: 32 months vs. 15 months, P=0.033), but this effect exists only in the SMARCA4-mutated group.

Currently, there are no targeted drugs directly against SMARCA4 mutations, and sensitivity to platinum-based chemotherapy is low. However, the high TMB signature suggests that some patients may benefit from immunotherapy combined with chemotherapy (e.g., the 5-year OS rate with camrelizumab combined with chemotherapy reached 27.8%). SMARCA4 mutation is associated with low PD-L1 expression and reduced CD8+ T-cell infiltration, but high TMB may suggest potential benefit from immunotherapy.

The ABCP regimen has a synergistic mechanism: Atezolizumab (anti-PD-L1): reverses the immunosuppressive microenvironment; Bevacizumab (anti-VEGF): inhibits angiogenesis and enhances T-cell infiltration; Platinum + Paclitaxel: directly kill tumor cells and release neoantigens. Therefore, the investigators preset that SMARCA4 mutation may affect chemotherapy/immunotherapy response through epigenetic regulation, and its value as a predictive biomarker needs to be validated. Hence, the purpose of this study is to observe and explore the efficacy and safety of first-line ABCP four-drug combination therapy in patients with advanced SMARCA4-mutated non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with pathologically confirmed NSCLC, meeting the following criteria based on the IASLC 9th Edition Lung Cancer TNM Staging System (International Association for the Study of Lung Cancer/Union for International Cancer Control): Histologically or cytologically confirmed unresectable locally advanced (Stage IIIB/IIIC) disease not amenable to curative-intent concurrent chemoradiotherapy, metastatic, or recurrent (Stage IV) non-squamous NSCLC;
2. Confirmed SMARCA4 mutation (verified by NGS testing);
3. ECOG performance status 0-1, with no prior systemic anticancer therapy;
4. Absence of driver gene mutations (e.g., EGFR, ALK, ROS1);
5. Patients capable of providing sufficient blood samples (detailed in sample requirements) and complete baseline clinical data, including: age, gender, smoking history, family history, lesion location(s), lesion size(s), number of lesions, tumor markers, pathological indicators, treatment records, and re-examination/follow-up information;
6. Voluntary participation with signed informed consent form, willingness to undergo follow-up assessments and provide treatment process details, efficacy data, and prognostic information, with commitment to complete the entire study.

Exclusion Criteria:

* (1) Active autoimmune diseases or interstitial lung disease; (2) Bleeding tendency or contraindications to Bevacizumab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Treatment-naive patients with advanced SMARCA4-mutated NSCLC
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2025-08-20 (Estimated); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | through study completion, an average of 1 year
  Objective Response Rate (ORR): Assessed according to RECIST v1.1 criteria to evaluate the antitumor activity of the ABCP regimen.
Progression-Free Survival | through study completion, an average of 1 year
  Progression-Free Survival (PFS): Defined as the time from enrollment to disease progression or death.

CONTACTS AND LOCATIONS:
Locations (1):
- The 900th Hospital of the Joint Logistic Support Force, PLA, Fuzhou, Fujian, China, 350025, Fuzhou, China

IPD SHARING:
Plan to Share IPD: No